CLINICAL TRIAL: NCT05106010
Title: The Effect of Yoga on Decreasing Risk of Fall-Related Injury in Peri and Post-Menopausal
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Cathy Arnold, Professor, University of Saskatchewan
Other Study IDs: Bio 17-64
Record Dates: First submitted 2021-08-25; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Fall Injury; Incontinence; Balance; Distorted

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual Activity: Participants continued with usual activity, not participating in any yoga intervention for 12 weeks
- Balance Flow Yoga: Community hatha yoga flow class, 75 minutes duration, twice per week for 12 weeks
  Interventions: Other: Balance Flow Yoga

INTERVENTIONS:
Other: Balance Flow Yoga — The yoga class is based on hatha yoga which includes physical poses and mindful movement integrated with breath. Conducted in a local yoga studio for 75 minutes duration, twice per week and also open to the public. The specific yoga techniques reflect the objectives of our study and focus on addressing some of the physical, mental and emotional factors that potentially contribute to falls such as balance, balance confidence, strength, coordination, proprioception, core training strategies, and breathing techniques integrated with mindfulness practices and yoga philosophy. The practices will incorporate a combination of seated, kneeling, standing and lying postures and transitions between positions with individual modifications provided on an as-needed basis. The yoga classes will be co-designed by registered yoga teachers and taught by two trained and experienced and yoga teachers blinded to study testing measures.
  Groups: Balance Flow Yoga

SUMMARY:
The primary objective of this study is to evaluate the effect of yoga on both fall risk factors AND capacity to successfully control landing and descent during a simulated fall among peri-and post- menopausal women. Older women are particularly vulnerable to sustaining fall-related injuries and although targeted exercises focusing on balance and strength may decrease the risk of falls, the ideal type of intervention to prevent injury when a fall is unavoidable is not known. Yoga is an increasingly popular health practice with potential benefits linked to improving balance, muscle strength and quality of life, but there is no evidence that yoga can improve the capacity to reduce the risk of fall-related injury. Such evidence will help to inform health promotion and fall/injury risk management for older adults.

DETAILED DESCRIPTION:
Falls are the leading cause of injury hospitalization for older adults in Canada. Determining effective and feasible community-based interventions is important to prevent the downward spiral of failing health, admission to long term care and even death following a serious fall-related injury. Women in their 50s and 60s are particularly vulnerable to sustaining fall-related injuries such as fractures. Our research team has identified early signs of fall risk in women aged 50 to 65 years. Exercise is known to decrease fall risk in community-dwelling older adults when components of balance, strength and agility are included, but the evidence is not clear on the effect of different types of exercise on decreasing fall-related injury risk particularly for older women at risk in their peri-menopausal and early post-menopausal years.

The risk of injury from falls depends on both the severity of impact and neuromuscular capacity such as bone and muscle strength of the affected body part. Most falls in community-dwelling older women occur in a forward direction. Forward falls are typically combined with hand contact as a protective response to prevent head, hip or torso injury. Evidence from the investigators' research team suggests that women in their 60s and 70s years do not have the same capacity to control a safe landing and decrease force impact compared to women in their 20s or 30s.Older women also demonstrate diminished activation of the abdominal core muscles prior to an unexpected simulated fall. The impact of diminished pelvic floor muscle control could also be a contributing factor to fall and injury risk in peri- and post-menopausal women as it has been associated with decreased balance, urinary incontinence and fall risk.

Yoga is a common recreational choice for peri- and post-menopausal women. Reasons could include a range of health improvements such as easing menopausal symptoms, improving pelvic floor dysfunctions such as incontinence or pelvic pain, enhancing bone loading to combat early osteoporosis, and improving overall quality of life. Yoga has also been associated with benefits to decrease fall risk; however, there is no substantive evidence that these outcomes result in a decrease in fall rates or a reduction in the injuries associated with falling.

Yoga, a system of health that promotes physical, mental, emotional, social and spiritual well-being, may offer unique benefits to decrease both fall risk and injury risk in the event a fall is unavoidable. Hatha yoga includes physical poses, mindful movement, breath awareness and regulation practices that can address balance, flexibility, and promote upper body loading and whole body strength training. The additional focus on abdominal and pelvic floor core control and breath techniques during functional movement may also promote motor control important in the maintenance of balance and enhance protective responses and landing strategies. The positive mental health focus and meditative component of linking physical postures and movement to breath could also help to improve balance confidence and decrease fear of falls. Yoga has multiple promising benefits to decrease the risk of fall-related injury in older women but there remains gaps in the literature to substantiate these claims.

The primary research questions are:

1. What is the effect of 12 weeks of hatha yoga on fall risk factors in peri- and post-menopausal women? (balance, balance confidence, functional mobility, muscle strength, incontinence leakage, symptoms and bother) and
2. Does 12 weeks of hatha yoga improve capacity to land and control the descent of a forward fall in peri- and post-menopausal women? (muscle activation, range of motion, reaction time, and energy absorption).

   Secondary research questions will explore:
3. What are the perceived changes in general health, fall risk, menopausal symptoms and incontinence for women who participate in yoga? What are the motivators, facilitators and barriers for participation in a regular yoga practice?

ELIGIBILITY:
Inclusion Criteria:

* women, age 50 to 70 years

Exclusion Criteria:

* participation in yoga twice per week or more in the past three months
* any recent upper extremity (UE), neck or back injury, or other painful joint problem that significantly limits day to day activities
* distal radius fracture in the past two years, any fracture in the past year, or a history of multiple fractures of the wrist or forearm
* any history of UE neurological problems (i.e. Stroke, Multiple Sclerosis, Parkinson's disease, reflex neuropathy)
* any cardio-vascular problems that would contradict maximum effort strength assessment
* presence of a joint replacement (i.e. hip or knee)
* unable to safely ambulate independently (with or without a walking aid) in the community.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self selected as female/woman
Study Population: Women age 50 to 70 years of age
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Muscle Strength Grip Change | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  Grip strength using a hand held dynamometer
Muscle Strength Shoulder and Elbow Change | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  Shoulder flexion, abduction and elbow extension using hand-held dynamometer
Muscle Strength Upper Body Change | 12 weeks
  concentric and eccentric upper body strength test using isokinetic dynamometer
Balance Change | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  mini-BESTest, comprehensive balance assessment of four balance systems
30 second chair stand change | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  number of sit to stand motions in 30 sec
one leg stand change | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  seconds standing on one leg, up to 60 sec
modified clinical test of sensory interaction and balance change | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  four balance conditions, maximum score = 120 seconds, meaning better balance
balance confidence change | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  activities balance confidence scale (ABC) maximum score 100 meaning higher confidence
incontinence-ICIQ-UI short form and FLUTS change | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  International Consultation on Incontinence Modular Questionnaire and the Urinary Incontinence short form; includes symptoms of bother, stress and urge. It is scored on a scale from 0-16 for symptoms of filling, 0-12 for voiding symptoms and 0-20 for incontinence symptoms
incontinence-pad test change | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  weight (grams) of pad pre and post water consumption and activity protocol
range of motion change | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  wrist extension and shoulder extension using goniometer (degrees)
kyphosis change | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  thoracic kyphosis index with flexicurve ruler (degrees)
reaction time | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  time (seconds) from hand motion to touching forceplate at shoulder level in standing
biomechanical outcomes landing on outstretched hand | change assessed 12 weeks after baseline, and after 12 weeks of intervention
  impact force, energy absorption, range of motion, torque in both controlled and unexpected descent in a simulated forward fall lab apparatus

SECONDARY OUTCOMES:
perceptions of experience | 24 weeks after baseline
  benefits, challenges and experiences determined from focus groups (qualitative)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
Requests can be made to PI